CLINICAL TRIAL: NCT05054660
Title: Applying a Chatbot to Geriatric Patients in Psychiatric Clinics: A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Taipei University of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202001915B0C601
Record Dates: First submitted 2021-09-01; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-08

CONDITIONS: Loneliness; Geriatric Depression
Keywords: geriatric psychiatry; chatbot; conversational agent

STUDY DESIGN:
Intervention Model Description: psychiatry outpatient using the investigator-developed-chatbot, and evaluate effectiveness, acceptability, usability, and adoption
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- caring chatbot (Experimental): The investigators will enroll participants aged over 55 in the psychiatric outpatient department. The participants will get a one-month caring chatbot and can interact with the chatbot freely.
  Interventions: Other: caring chatbot

INTERVENTIONS:
Other: caring chatbot — The investigators will use the developed caring chatbot to provide care to the cases and to collect case treatment data and interaction data between the case and the caring chatbot.

SUMMARY:
This study will use the caring chatbot developed by the Taipei University of Technology team to provide care for participants and use robots to talk to them to collect daily changes in mood, sleep, and activities, and analyze the factors that affect the physical and mental health of the elderly.

DETAILED DESCRIPTION:
The prevalence of anxiety and depression in middle-aged and elderly people is quite high. Among the risk factors for illness, "loneliness" is closely related to the physical and mental health of the elderly: the higher the loneliness of the elderly, the more likely to develop unhealthy lifestyle habits and emotional symptoms such as depression and anxiety. Depression and anxiety are often comorbid, and the diagnoses of the two groups have many symptoms that overlap each other. Emotional symptoms that have not been effectively treated have a great impact on the quality of life, and the drug treatment of emotional disorders in the elderly is more difficult. In addition to medication, maintaining a healthy lifestyle is also conducive to the control of emotional disorders.

Information technology has been used in supplementary medical care and maintenance of physical and mental health for decades. However, reviewing the literature, there is less research on applications developed in cooperation between the information field and the field of psychiatric medical care, and there are no applications developed for the mental health of middle-aged and elderly people.

This study will use the caring chatbot developed by the National Taipei University of Technology team to provide care for the participants enrolled from the psychiatric outpatient department, and use the chatbot to talk to them to collect daily changes in mood, sleep, and activities, and analyze the factors that affect the mental health of the elderly.

This research anticipates the following goals:

1. With the chatbot developed, it provides care for subjects every day and collects their daily changes in mood, sleep, and activities.
2. Analyze the relationship between robot interaction and emotional changes, and evaluate the impact of chatbot intervention on the health behavior of the case.

ELIGIBILITY:
Inclusion Criteria:

* with the diagnosis of persistent depressive disorder, major depressive disorder, general anxiety disorder, panic disorder, or agoraphobia
* the condition of their disease is relatively stable (defined as no thought of death and no medication adjustment in the recent 3 months).
* Have a personal mobile phone or communicator that can connect to the Internet

Exclusion Criteria:

* Those who are unwilling to participate in this research
* Those who have poor assessment ability by clinicians and cannot understand the content of the questionnaire; or those who cannot continue to complete the test due to their physical condition
* Comorbid schizophrenia or bipolar disorder
* Patients with dementia, brain injury, substance abuse, and stroke

Ages: 55 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-09-27 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
acceptance measured by seven-point Likert scales | at the end of one-month-intervention of the caring chatbot
  Satisfacation (How satisfied were you with Chatbot?), usability (How easy was talking to Chatbot?), continue (How much would you like to continue working with Chatbot?) and adherence (How likely is it that you will follow Chatbot's advice?) were measured by single items on seven-point Likert scales (with 1= "not at all" and 7="very much").

SECONDARY OUTCOMES:
Change from baseline "loneliness" measured by UCLA Loneliness Scale | before and at the end of one-month-intervention of the caring chatbot
  The UCLA Loneliness Scale (version 3) is a 20-item measure that assesses how often a person feels disconnected from others. Using a 4-point rating scale (1= never; 4 = always), participants answer 20 questions, and researchers later reverse-code the positively worded items so that high values mean more loneliness.
Change from baseline "depression" measured by Geriatric Depression Scale-Short Form (GDS-15) | before and at the end of one-month-intervention of the caring chatbot
  Geriatric Depression Scale (GDS) is designed for the older population. A Short Form GDS consisting of 15 questions. Of the 15 items, 10 indicated the presence of depression when answered positively, while the rest indicated depression when answered negatively. Scores of 5-8 indicate mild depression; 9-11 indicate moderate depression; 12-15 indicate severe depression.
Change from baseline "anxiety" measured by Hospital Anxiety and Depression Scale- Anxiety subscale | before and at the end of one-month-intervention of the caring chatbot
  Hospital Anxiety and Depression Scale (HADS) is developed for people with physical illnesses. This scale includes a total of 14 questions. There are 7 questions about anxiety and depression, each with a 4-point scoring method (0-3 points). The higher the total score, the greater the anxiety or the greater the depression. Due to the high overlap between the topics of the depression subscale and the GDS, this study only uses the anxiety subscale.
Change from baseline "quality of life" measured by Short Form Quality Life Sale (SF-12) | before and at the end of one-month-intervention of the caring chatbot
  Short Form Quality Life Sale (SF-12) is the most commonly used questionnaire in the study of the quality of life of the elderly, with a total score ranging from 13~43. A higher score reflects a better life quality.
Change from baseline "physical activity" measured by International Physical Activity Questionnaire Self-Administered Short Version (IPAQ-SS) | before and at the end of one-month-intervention of the caring chatbot
  International Physical Activity Questionnaire Self-Administered Short Version (IPAQ-SS) measures the physical activity of the participant in the past seven days by self-filled method. The questionnaire is consisted of four domains: (1)during transportation, (2) at work, (3) during household and gardening tasks and (4) during leisure time, including exercise and sport participation. In each of the four domains the number of days per week and time per day spent in both moderate and vigorous activity are recorded.